CLINICAL TRIAL: NCT02140710
Title: The Impact of Visceral Osteopathic Treatment on the Meconium Evacuation in Very Low Birth Weight Infants
Brief Title: Impact of Visceral Osteopathic Treatment on Meconium Evacuation in Preterm Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Nadja Haiden,MD, M.D., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OST2010
Record Dates: First submitted 2014-05-10; First posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Meconium Ileus
Keywords: premature infant; visceral osteopathy; alternative medicine; meconium passage; enteral feedings; hospital stay
MeSH Terms: conditions — Meconium Ileus; Premature Birth | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Osteopathic treatment group (Active Comparator): visceral osteopathic treatment algorithm
  Interventions: Procedure: Osteopathic treatment
- Control group (No Intervention): no intervention

INTERVENTIONS:
Procedure: Osteopathic treatment — visceral osteopathic treatment algorithm: Global listening and local listening on the abdomen Release lower ribs and thoracic diaphragm Pylorusrelaxation Release of the Duodenum and the C-Loop Small intestine diagnosis- Lifting the gut and bringing it to a stillpoint Root of mesentery diagnosis (and manipulation) Mobilisation of the ileocoecalic valve Mobilisation of colon ascendens, transversum, descendens Root of sigmoid diagnosis and manipulation
  Arms: Osteopathic treatment group

SUMMARY:
Timing of the first and last meconium stool is critical for oral feeding tolerance and proper gastrointestinal function. The time until premature infants pass their first meconium ranges from 1 hour to 27 days (median: 43 hours). Obstruction of the gastrointestinal tract by tenacious, sticky meconium frequently leads to gastric residuals, a distended abdomen and delayed food passage Recent data support the concept that complete rapid evacuation of meconium plays a key role in feeding tolerance . If duration to full enteral feedings is extended, the probability to acquire infections due to intravenous access for parenteral nutrition increases and hospital stay of the infant prolongates. Previously two prospective trials focusing on the problem of delayed meconium evacuation in preterm with different therapeutic pharmacological approaches were published by our group. None of the applied therapies appeared to be effective or had a beneficial effect- quite the contrary one agent (Gastrografin) was supposed to have severe negative side effects. Therefore we were looking for an alternative, non-invasive, holistic solution for the problem of delayed meconium excretion. Osteopathic treatment with the emphasis on the relationship of the structural and functional integrity of the body and with its variety of therapeutic manual techniques seemed to be remedy. Treating the abdomen of premature infants with visceral osteopathic techniques might be more effective to mobilize meconium from small bowel and deep parts of the colon. Therefore we hypothesized that repeated visceral osteopathic treatment accelerates meconium evacuation in premature infants, and thereby enhances feeding tolerance in this population.

ELIGIBILITY:
Inclusion Criteria:

* premature infants with a birthweight 1500 gram

Exclusion Criteria:

* major congenital malformations
* known gastrointestinal abnormalities

Ages: 60 Minutes to 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
complete meconium evacuation | days up to 100 days of life
  Primary outcome parameter was specified as complete meconium excretion. The time to complete meconium evacuation was defined as day of life on which the last meconium was passed. The nursing staff assessed the quality of stools as "meconium" (black, thick, sticky) or "non meconium" by appearance and documented data into the electronic patient documentation system.

SECONDARY OUTCOMES:
Time to full enteral feedings | days up to 100 days of life
Introduction of enteral feedings | days up to 100 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Haiden, M.D., Principal Investigator — MUV
Locations (1):
- Nadja Haiden, Vienna, Austria

REFERENCES:
- [Derived] Haiden N, Pimpel B, Kreissl A, Jilma B, Berger A. Does visceral osteopathic treatment accelerate meconium passage in very low birth weight infants?- A prospective randomized controlled trial. PLoS One. 2015 Apr 15;10(4):e0123530. doi: 10.1371/journal.pone.0123530. eCollection 2015. PMID 25875011